CLINICAL TRIAL: NCT03335189
Title: Adaptation, Feasibility and Acceptability Study of the Advanced Symptom Management System (ASyMS) Mobile Health Intervention to Reduce Chemotherapy Toxicities in Canadian Cancer Patients
Brief Title: Feasibility Study of the Advanced Symptom Management System (ASyMS) in Canadian Cancer Patients
Acronym: ASyMS-Can
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CAPCR ID: 17-5367.0
Record Dates: First submitted 2017-10-17; First posted 2017-11-07 (Actual); Last update posted 2019-06-07 (Actual); Status verified 2019-06

CONDITIONS: Supportive Care; Cancer
Keywords: E-Health; Smartphone technology; Real-time symptom assessment; Self-care; Symptom management
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ASyMS-Can (Experimental): TParticipants assigned to the experimental group will be provided with the encrypted, secure, pre-programmed ASyMS-Can android phone, and instructed of its use; how to report their symptomatology on a twice daily basis using the CTAQ for the first 14 days of each treatment cycle until end of the final cycle of treatment (or up to 16 weeks).
  Interventions: Device: ASyMS-Can
- Control (No Intervention): Control group will be asked to complete the study questionnaires at your clinic visits. Also, research staff will contact participants at 1 to 14 days following each chemotherapy, mid and end of each chemotherapy appointment and again within week 8 and 16 of your participation to collect information about participants' symptoms.

INTERVENTIONS:
Device: ASyMS-Can — Data reported by the participants will be sent to a secure, encrypted clinical central server hosting the risk-alerting algorithms. The web interfaces will provide a clinical portal for the nurses to screen and follow any alerts being triggered, as well as review patient-specific information. Based on these back-end computations, participants will receive automated self-care notifications on their mobile phones. If incoming symptom reports indicate severe adverse effects a designated clinic nurse will receive an 'amber alert', or 'red alert', that will require response within 30 minutes. Nurses will handle alerts during business hours (9 am to 5 pm). After-hour alerts will be sent to the oncologist or nursing supervisor on call as per usual care. Patients will be instructed that clinicians will not receive alerts during the evening hours or night and instructed to follow usual practice of contacting their family physician, or oncologist on call, or call 911, as required.
  Other Names: ASyMS
  Arms: ASyMS-Can

SUMMARY:
The Advanced Symptom Monitoring and Management System - Canada (ASyMS-Can) is a remote phone-based symptom management system that prompts patient self-care and clinician telephone triage and intervention based on alerts for managing cancer treatment side effects such as nausea and vomiting, fatigue, etc. ASyMS-Can is an android phone-based application that is given to patients to self-report their symptoms using a patient reported outcome symptom questionnaire and level of severity daily, on a secure mobile android phone, from home or outside of clinics. Based on back-end computations, patients receive automated self-care notifications on their mobile phones with advice on self-care for mild to moderate severe symptoms. The system also in the case of severe symptoms will alert the designated clinic nurse to prompt electronic telephone triage and intervention (yellow alert response in 4 hours or within 30 minutes for severe symptoms-red alert).

DETAILED DESCRIPTION:
In addition, patients can access a self-care library and symptom graphs (detailing trends in individual symptoms experienced) through the ASyMS-Can patient phones. If the incoming symptom reports are of clinical concern, the server software will generate two levels of alerts (amber& red) that will be sent to the designated nurse, who will receive alerts on a dedicated ASyMS-Can nurse handset (mobile phone). The nurse will view the patient's symptom reports on a secure web page, and contact the patient directly at home by telephone, guided through a decision-support algorithm on the web-based platform to systematize the triage based on the COSTARS guideline, facilitating the initiation of "real-time" clinical interventions. An "amber alert", which requires response within 4 hours, indicates that the symptom(s) are not severe or life-threatening but early intervention might prevent further symptom progression. The second level of the triage alert, 'red alert', will be sent to the nurse for severe symptoms and will require response within 30 minutes of receipt of the alert

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with early stage breast, colorectal, and lymphoma (Hodgkin's [HD], non- Hodgkin's [NHL].
2. Scheduled to receive 2-, 3- or 4-weekly chemotherapy protocols (i.e. chemotherapy administered at repeated cycles of 14, 21 or 28 days, respectively).
3. Scheduled to receive a minimum of 3 cycles of systemic chemotherapy (any regimen); adjuvant or neo-adjuvant on an out-patient basis;
4. Adults >=18 years of age;
5. Able to provide written consent and willing to participate;
6. Adequate ability to use or be trained in use of a mobile phone for symptom reporting

Exclusion Criteria:

1. Enrolled/receiving an investigational treatment;
2. Scheduled to receive concurrent radiotherapy during chemotherapy treatment.
3. Scheduled to receive weekly chemotherapy protocols. In addition, patients who shift from a 2-, 3- or 4-weekly protocol to a weekly protocol during chemotherapy will be excluded from further participation in the study.
4. Any distant metastasis based on Ann Arbor or TNM staging
5. Unable to speak/read/write English sufficiently to complete study measures.
6. Unable to complete study measures due to a pre-existing disability (e.g. visually impaired)
7. Cognitive impairment/severe pre-existing emotional issues as assessed by the treatment team which may impede completion of study measures.
8. Low performance status (ECOG > or =3)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-05-28 (Actual)

PRIMARY OUTCOMES:
Feasibility of recruitment | Recruitment rate aim is 7-8 patients/month, for 1 year.
  Recruitment Rate (RRa)

SECONDARY OUTCOMES:
Symptom Severity | Baseline (within 1 week before 1st chemotherapy cycle). Mid-way each chemotherapy cycle, (Day 6-8, 9-11, or 13-15 - dependent on number of days in the chemotherapy cycle).
  Symptom severity will be measured using the Memorial Symptom Assessment Scale (MSAS). The MSAS is a multidimensional self-report questionnaire that evaluates 32 physical and psychological symptoms according to their frequency, severity and distress/bother to the person in the past week.
Chemotherapy Self-Management Behaviours | Midpoint of treatment cycle (Week 3-4, or 7-8 - dependent on chemotherapy regimen being given).
  Chemotherapy Self-Management Behaviours will be measured using the Leuven questionnaire for self-care behaviours during chemotherapy (L-PaSC). The L-PaSC is a 22-item instrument with 7 themes that capture the most relevant aspects of patient self-care during chemotherapy.
Self-Efficacy for Coping | Baseline (within 1 week before 1st chemotherapy cycle), midpoint of treatment cycle (Week 3-4, or 7-8 - dependent on chemotherapy regimen being given), and end of treatment (Week 6-8 or 14-16-dependent on chemotherapy regimen being given).
  Self-efficacy will be measured using the Cancer Behavior Inventory (CBI-B) which is a 12-item unidimensional instrument designed to assess coping self-efficacy of cancer patients.
Psychological Distress | Baseline(within 1 week before 1st chemotherapy cycle), midpoint of treatment cycle (Week 3-4, or 7-8 - dependent on chemotherapy regimen being given), and end of treatment (Week 6-8 or 14-16-dependent on chemotherapy regimen being given).
  Using the Depression, Anxiety and Stress Scale (DASS21) which contains 21 items for self-reporting for measuring a range of symptoms common to both depression and anxiety. Each item is scored from 0 (did not apply to me at all over the last week) to 3 (applied to me very much for most of the time over the past week).
Information and Support Needs | Baseline(within 1 week before 1st chemotherapy cycle), midpoint of treatment cycle (Week 3-4, or 7-8 - dependent on chemotherapy regimen being given).
  Using the Cancer Treatment Scale (CaTS) that is a two factor, 25-item measure that assesses sensory/psychological concerns and procedural concerns relating to cancer treatment.
Health Related Quality of Life | Baseline(within 1 week before 1st chemotherapy cycle), midpoint of treatment cycle (Week 3-4, or 7-8 - dependent on chemotherapy regimen being given), and end of treatment (Week 6-8 or 14-16-dependent on chemotherapy regimen being given).
  EuroQual-5D-5L (EQ-5D-5L). The questionnaire offers 5 levels of response for 5 dimensions including Mobility, Self-care, Usual Activities, Pain/Discomfort, and Anxiety/Depression.
Health Service Utilization | End of each chemotherapy cycle (Week 2-3, or 4-5 - dependent on chemotherapy regimen being given).
  Including days in hospital, ED visits, urgent care use, unscheduled clinic visits) self-reported by patients at end of each treatment cycle and calculated as group proportions over the entire course of treatment.
Acceptance, Patient User/Satisfaction, System Usefulness, Information Quality and Interface Quality of User Interface | End of study (Week 16)
  Using the Post-Study System Usability Questionnaire (PSSUQ) that consists of 16 items which produce four scores-one overall and three sub-scales. The questionnaire designed to assess users' perceived satisfaction with computer systems or applications. The self-administered questionnaire are composed of multiple separate items organized into scales, with each scale assumed to measure an attribute or attitude dimension is a common approach to usability evaluation.
Clinicians' acceptance | End of study (Week 16)
  using the Treatment Evaluation Inventory Short-Form (TEI-SF)

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Moradian S, Krzyzanowska M, Maguire R, Kukreti V, Amir E, Morita PP, Liu G, Howell D. Feasibility randomised controlled trial of remote symptom chemotherapy toxicity monitoring using the Canadian adapted Advanced Symptom Management System (ASyMS-Can): a study protocol. BMJ Open. 2020 Jun 17;10(6):e035648. doi: 10.1136/bmjopen-2019-035648. PMID 32554724